CLINICAL TRIAL: NCT03990259
Title: Penyagolosa Trail Saludable Women
Acronym: PTSW
Status: Completed | Type: Observational
Sponsor: Universitat Jaume I (Other)
Collaborators: Club Deportivo Marató i Mitja Castelló-Penyagolosa (Unknown); Fundación Vithas-Nisa (Unknown); Hospital Vithas-Nisa 9 de Octubre (Unknown)
Responsible Party: Sponsor
Other Study IDs: UJI_PTSW001
Record Dates: First submitted 2019-05-20; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Physical Exertion
Keywords: Ultraendurance; Sex differences; Performance; Genetics; Physiological damage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — The genomic DNA was isolated from a saliva sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male: The male individuals of the study population
  Interventions: Other: Running the CSP Mountain Race
- Female: The female individuals of the study population
  Interventions: Other: Running the CSP Mountain Race

INTERVENTIONS:
Other: Running the CSP Mountain Race — The runners completed a 107,6 km mountain race

SUMMARY:
This study has as main objective to asses different genetic, biochemical and physiological biomarkers affecting performance and health status in ultraendurance runners according to individual's sex.

DETAILED DESCRIPTION:
Ultraendurance races has been shown to impact on several health-related biomarkers, and therefore they may have detrimental effects on runners' health. In this study, we aim to analyze the impact of running a 107,6 km mountain race in ultraendurance runners splitting our sample by individual's sex.

To do this, baseline measurements of the runners have been collected through stress tests and biochemical analyses of blood and urine samples. Indeed, a saliva sample was collected to isolated a genomic DNA sample of each runner.

During the race anthropometrical, ventilatory and strength data was collected in three different moments and after crossing the finish line. Indeed, after completed the ultraendurance mountain race, blood and urine samples were taken at the finish line, as well as 24h and 48h post-race.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (>18 years old)
* Volunteers should be finish at least one ultraendurance mountain race (>60km).

Exclusion Criteria:

* Having heart disease
* Having kidney disease
* Taking a medication on an ongoing basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 ultraendurance amateur runners, 19 females and 31 males.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Change in the biochemical parameters related to kidney injury, dehydration, inflammation, and cardiac damage | 12 hours before the race, 15 minutes after the race, 24 hours after the race and 48 hours after the race
  Blood concentration of estradiol, testosterone, progesterone, creatinine, troponin, C-reactive protein, hemoglobin, sodium, potassium, chlorine, iron, and ferritin. Concentration of all these parameters is expressed in mass per volume (i.e. nanograms per milliliter)
Change in the biochemical parameters related to muscle damage | 12 hours before the race, 15 minutes after the race, 24 hours after the race and 48 hours after the race
  Blood concentration of lactate dehydrogenase and creatine kinase. The enzyme concentration is expressed in units per volume (enzyme units per milliliter)
Change in the biochemical parameters related to immunological response | 12 hours before the race, 15 minutes after the race, 24 hours after the race and 48 hours after the race
  Blood concentration of erythrocytes, hematocrit, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and platelet volume. The concentration of each cell type is expressed in number of cells per volume (cells per liter)
Change in the power level | 12 hours before the race, 15 minutes after the race
  Squat Jump (high of the jump measured in centimeters)
Change in the lung function | 12 hours before the race, and 15 minutes after the race
  Pulmonary function test by spirometry. The parameters measured are vital capacity (VC), forced vital capacity (FVC), maximal mid-expiratory flow (MEF) and total lung capacity. Outcome data of all these parameters are expressed in liters.
Change in the lung function related to time | 12 hours before the race, and 15 minutes after the race
  Pulmonary function test by spirometry. The parameters measured are forced expiratory volume in 1 second (FEV1) and in 6 seconds (FEV6) and peak expiratory flow (PEF). Outcome data of all these parameters are expressed in liters per second.
Change in the Strength level | 12 hours before the race, in three moments during the race (after running 33km, 65km and 94 km), and 15 minutes after the race
  Hand grip (pressure in kilograms)
Change in the Ventilatory Flow | 60 minutes before the race, in three moments during the race (after running 33km, 65km and 94 km), and 15 minutes after the race
  Ventilatory Flow measurement (liters per minute)
Change in the biochemical parameters related to dehydration and kidney injury | 60 minutes before the race and 15 minutes after the race
  Urine test to measure the concentration of sodium and creatinine, as well as urine density
Analysis of tne changes in the Physical activity data | From 9 hours before starting the race to 48 hours after crossing the finish line.
  Physical activity measured by wearing accelerometer devices. Physical activity defined as sedentary, light, moderate, vigorous, very vigorous and extremely vigorous. The aim to wear accelerometers devices is to monitor individuals.
Analysis of the presence or absence of genetic markers related to endurance performance and ability to muscle damage recovery | 12 hours before the race
  Analysis of different polymorphisms in genomic DNA samples, which were isolated from the saliva sample of each participant.
Telomere length, genetic marker related to biological aging | 12 hours before the race
  Analysis of the telomere length in genomic DNA samples, which were isolated from saliva samples of each participant

SECONDARY OUTCOMES:
Self-reported questionnaire about social and health status | One month before the race day
  Personal questionnaire asking for social status. Multiple-choice questions. Participants choose one of the different possible answers. Data is encoded as a factor variable with different levels.
Self-reported questionnaire about training habits | One month before the race day
  Personal questionnaire asking for training habits. Multiple-choice questions. Participants choose one of the different possible answers. Data is encoded as a factor variable with different levels.
Self-reported questionnaire about menstrual cycle (only for females) | One month before the race day
  Personal questionnaire asking for training habits. Open-ended questions. Females answer questions regarding menstrual cycle (duration, dates, regularity, quantity of bleeding, pregnancy history, dysmenorrhea).
Assesment of physical condition by cardiopulmonary test | One month before the race day
  Maximal oxygen consumption (milliliters of oxygen used in one minute per kilogram of body weight)
Analysis of body composition (proportion of body fat, fat-free mass and water) per body areas (trunk, arms and legs) | 12 hours before the race, and 15 minutes after the race,
  Bioimpedance analysis (percentage of body fat, fat-free mass and water)
Heart rate | Through race completion (the time that a runner is performing the 107 kilometers of the race, an average of 25 hours)
  Recording the number of contractions of the heart per minute (bpm) by using a heart rate monitor during the race
Evaluation of effort subjective perception | 60 minutes before the race, in three moments during the race (after running 33km, 65km and 94 km), and 15 minutes after the race
  Borg ratings of perceived exertion (CR10). Scale with ten levels (0-Nothing at all, and 10-Extremely)
Evaluation of muscle damage subjective perception per body areas | 12 hours before the race, 15 minutes after the race, and 48 hours after the race
  Evaluation of perceived muscle damage in a 10-level scale. Scale with ten levels (0-Nothing at all, and 10-Extremely)
Change in the body mass | 60 minutes before the race, in three moments during the race (after running 33km, 65km and 94 km), and 15 minutes after the race,
  Body mass measurement (weight in kilograms)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hernando, PhD, Principal Investigator — Universitat Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No
It is not planned to share participant's data

REFERENCES:
- [Background] Cheuvront SN, Carter R, Deruisseau KC, Moffatt RJ. Running performance differences between men and women:an update. Sports Med. 2005;35(12):1017-24. doi: 10.2165/00007256-200535120-00002. PMID 16336006
- [Background] Eichenberger E, Knechtle B, Rust CA, Rosemann T, Lepers R. Age and sex interactions in mountain ultramarathon running - the Swiss Alpine Marathon. Open Access J Sports Med. 2012 Jul 31;3:73-80. doi: 10.2147/OAJSM.S33836. eCollection 2012. PMID 24198590
- [Background] Gimenez P, Kerherve H, Messonnier LA, Feasson L, Millet GY. Changes in the energy cost of running during a 24-h treadmill exercise. Med Sci Sports Exerc. 2013 Sep;45(9):1807-13. doi: 10.1249/MSS.0b013e318292c0ec. PMID 23524515
- [Background] Hernando C, Hernando C, Collado EJ, Panizo N, Martinez-Navarro I, Hernando B. Establishing cut-points for physical activity classification using triaxial accelerometer in middle-aged recreational marathoners. PLoS One. 2018 Aug 29;13(8):e0202815. doi: 10.1371/journal.pone.0202815. eCollection 2018. PMID 30157271
- [Background] Joyner MJ. Physiological limits to endurance exercise performance: influence of sex. J Physiol. 2017 May 1;595(9):2949-2954. doi: 10.1113/JP272268. Epub 2017 Feb 9. PMID 28028816
- [Background] Knechtle B, Knechtle P, Rosemann T, Lepers R. Personal best marathon time and longest training run, not anthropometry, predict performance in recreational 24-hour ultrarunners. J Strength Cond Res. 2011 Aug;25(8):2212-8. doi: 10.1519/JSC.0b013e3181f6b0c7. PMID 21642857
- [Background] Knechtle B, Knechtle P, Wirth A, Alexander Rust C, Rosemann T. A faster running speed is associated with a greater body weight loss in 100-km ultra-marathoners. J Sports Sci. 2012;30(11):1131-40. doi: 10.1080/02640414.2012.692479. Epub 2012 Jun 6. PMID 22668199
- [Background] Ahmetov I, Kulemin N, Popov D, Naumov V, Akimov E, Bravy Y, Egorova E, Galeeva A, Generozov E, Kostryukova E, Larin A, Mustafina Lj, Ospanova E, Pavlenko A, Starnes L, Zmijewski P, Alexeev D, Vinogradova O, Govorun V. Genome-wide association study identifies three novel genetic markers associated with elite endurance performance. Biol Sport. 2015 Mar;32(1):3-9. doi: 10.5604/20831862.1124568. Epub 2014 Oct 21. PMID 25729143
- [Background] Borghini A, Giardini G, Tonacci A, Mastorci F, Mercuri A, Mrakic-Sposta S, Moretti S, Andreassi MG, Pratali L. Chronic and acute effects of endurance training on telomere length. Mutagenesis. 2015 Sep;30(5):711-6. doi: 10.1093/mutage/gev038. Epub 2015 May 22. PMID 26001753
- [Derived] Martinez-Navarro I, Aparicio I, Priego-Quesada JI, Perez-Soriano P, Collado E, Hernando B, Hernando C. Effects of wearing a full body compression garment during recovery from an ultra-trail race. Eur J Sport Sci. 2021 Jun;21(6):811-818. doi: 10.1080/17461391.2020.1783369. Epub 2020 Jun 30. PMID 32538286